CLINICAL TRIAL: NCT04992364
Title: Relationship Between Burnout Score and Clinical Performance on Anesthesiology and Intensive Therapy Residents
Brief Title: Clinical Impacts of Burnout Syndrome Among Anesthesiology Residents
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Doctor, Indonesia University
Other Study IDs: IndonesiaUAnes107
Record Dates: First submitted 2021-07-13; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Burnout, Caregiver
Keywords: anesthesiology; burnout; clinical performances; residency
MeSH Terms: conditions — Caregiver Burden; Burnout, Psychological

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive Clinical Performances: Subjects show positive clinical performances regarding burnout syndrome
  Interventions: Other: Burnout and Clinical performances questionnaires
- Negative Clinical Performances: Subjects show negative clinical performances regarding burnout syndrome
  Interventions: Other: Burnout and Clinical performances questionnaires

INTERVENTIONS:
Other: Burnout and Clinical performances questionnaires — Subjects were given questionnaires to assess burnout score and clinical performances

SUMMARY:
This study aimed to determine the relationship between burnout levels and clinical performances of anesthesiology residents.

DETAILED DESCRIPTION:
Fifty-five second until fourth year anesthesiology residents, who were not on any mental medication treatment, were recruited consecutively and asked to fill out questionnaires which are; the Maslach Burnout Inventory (MBI) questionnaire to assess burnout levels, Best Practice Anesthesiologist questionnaire to assess positive clinical performance, Anesthesiology Residents' Self-Reported Errors and Quality of Care questionnaire to assess negative clinical performance.

ELIGIBILITY:
Inclusion Criteria:

* second until fourth year anesthesiology residents
* not on any mental medication treatment
* willing to participate

Exclusion Criteria:

* on paid leave
* rejected to become the sample
* had their shift in 24 hours prior to this study

Ages: 25 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Anesthesiology residents who were on second until fourth year of residency
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Positive clinical performance | 1 month through study completion
  Subjects show positive clinical performance

SECONDARY OUTCOMES:
Negative clinical performance | 1 month through study completion
  Subjects show negative clinical performance

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided